CLINICAL TRIAL: NCT03506529
Title: Identification of Predictive Factors for Physiological Hypermetabolism of the Anal Canal in 18F-FDG PET / CT
Acronym: HYPHYCA
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03545-48
Record Dates: First submitted 2018-04-12; First posted 2018-04-24 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Anal Cancer
Keywords: TEP; hypermetabolism
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnary — questionnary on predictif factors about physiological hypermetabolism of anal canal

SUMMARY:
Questionnaire to be completed by patients coming for PET to identify the predictive factors of physiological hypermetabolism of the anal canal

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old
* Patient referred for 18F-FDG PET

Exclusion Criteria:

* History of surgery or anal and / or perineal and / or pelvic radiotherapy, whatever the indication
* Patient deprived of liberty, under tutorship or curatorship
* Any associated socio-educational, medical or psychological condition that could compromise the patient's ability to participate in the study (eg illiteracy, mental retardation, etc.)
* Pregnant woman (classic contraindication of a PET scan)
* Opposition of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient coming for a PET
Sampling Method: Non-Probability Sample
Enrollment: 644 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Description of predictive factors for physiological hypermetabolism of the anal canal in 18F-FDG PET / CT | Only at the day of inclusion, during an appointment for a TEP exam
  Confrontation in participants of hypermetabolism of the anal canal in PET with:
  number of stool/day and consistency of stool, medical history (by Answers to the specific questionnaire designed for the study)
PET analysis of hypermetabolism of the anal canal | Only at the day of inclusion, during an appointment for a TEP exam
  Visual analysis of hypermetabolism of the anal canal on a 3-point scale:
  0: no hypermetabolism
  1. moderate hypermetabolism
  2. intense hypermetabolism
CT scan with measurement | Only at the day of inclusion, during an appointment for a TEP exam
  measurement of the largest rectal diameter in mm.
CT scan with measurement | Only at the day of inclusion, during an appointment for a TEP exam
  Visual assessment of the rectal capacity on a 3-point scale (0, 1, 2) and content characteristics (air, feces, air and feces).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Caen
  - Centre François Baclesse, Caen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aide N, Tainturier LE, Nganoa C, Houdu B, Kammerer J, Galais MP, Ciappuccini R, Lasnon C. HYPHYCA: a prospective study in 613 patients conducting a comprehensive analysis for predictive factors of physiological 18F-FDG anal uptake. EJNMMI Res. 2020 Mar 20;10(1):28. doi: 10.1186/s13550-020-0615-5. PMID 32193623